CLINICAL TRIAL: NCT01920321
Title: Lung Volume Reduction in COPD Patients With an Inhomogeneous Severe Emphysema Located in the Upper Lobes, by Injecting Warm Saline Through the Bronchoscope Channel
Brief Title: Bronchoscopic Thermal Saline Ablation (BTSA) of Emphysematous Lung. A New Emphysema Therapy
Acronym: BTSA
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 195/12
Record Dates: First submitted 2013-07-16; First posted 2013-08-12 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Emphysema
Keywords: COPD; Bronchoscopic LVR; Emphysema; Hot injury
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endoscopic lung volume reduction (Experimental): After usual sedation, bronchoscope is introduce to the lung and palced in segmental wedge position then hot salineis instilled. Same procedure to others affected segments.
  Interventions: Procedure: Endoscopic lung volume reduction

INTERVENTIONS:
Procedure: Endoscopic lung volume reduction — Prior the procedure patients undergo - high resolution chest CT , extensive phisiological assessment.

SUMMARY:
Aim: To evaluate feasibility, safety and efficacy of relatively simple approach of bronchoscopic lung volume reduction (LVR) technology, independent of collateral ventilation.

Description: Patients with severe upper lobes heterogeneous emphysema, undergo unilateral bronchoscopic installation of saline thermal energy 50-55 ºC intending to induce an inflammatory airway and parenchymal injury and consequently fibrotic response resulting in LVR;

DETAILED DESCRIPTION:
Inclusion criteria:

1. Age 40-75 unlimited sex. 20 subjects
2. chronic obstructive pulmonary disease (COPD), GOLD 3-4 (global obstructive lung disease).
3. CT scan of lung and included high resolution slices. Demonstrating emphysematous, bullotic changes in the upper lobes.
4. Pulmonary function tests results- total lung capacity(TLC)>110%, residual volume(RV)>150%, diffusion of lung CO(DLCO)<80%,forced expiratory volume 1 second(FEV1):15-45%.
5. 6 minute walking distance (6MWD)> 140 meters.

Exclusion criteria:

1. Active ischemic heart disease, significant arrhythmia. ejection fraction (EF) <40%.
2. COPD that cause carbon bioxide(CO2) retention above 50 mm Hg and / or oxygen saturation at rest below 88%.
3. Pulmonary hypertension> 45 mmHg, according to the Echo Test.
4. . Cancer treatment with chemotherapy / radiation or expected life expectancy of less than two years.5. Pregnancy.

Methods: . A. Patient preparation and sedation as in diagnostic bronchoscopy. Sedation will be based on midzoln + demerol. The patients will be treated prior the treatment with Inhalation with salbutamol ans ipratropium bromide. Flexible bronchoscope with outer diameter 5 mm is introduced to the targated upper lobe, and placed in wedged position. This is followed by installion of 0.9% natriu, chloride(NaCl) at a temperature of 55ºC exit temperature 50ºC) in portions of 40 ml to 200 ml (in bronchoalveolar lavage up to 300 ml is acceptable. The patient is placed in horizontal position, and continuous ECG blood pressure. Oxygen saturation are monitored. This monitoring will be continue at least 2 hours after treatment. A chest x-ray is followed and the patient remain in the department for overnight.

Tracking: Minimum of 6 months - Outpatient follow up include in addition to physical examination extended pulmonary function test and after 3-6 months. low radiation chest CT.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-75 unlimited sex. 20 subjects
2. COPD, GOLD 3-4 (global obstructive lung disease).
3. CT scan of lung and included high resolution slices. Demonstrating emphysematous, bullotic changes in the upper lobes.
4. Pulmonary function tests results- TLC> 110%, RV> 150%, DLCO <80%,FEV1: 15-45%.
5. 6 minute walking distance > 140 meters.

   -

Exclusion Criteria:

1. Active ischemic heart disease, significant arrhythmia. Ejection fraction (EF) <40%.
2. Chronic lung disease that cause CO2 retention above 50 mm Hg and / or oxygen saturation at rest below 88%.
3. Pulmonary hypertension> 45 mmHg, according to the Echo Test.
4. . Cancer treatment with chemotherapy / radiation or expected life expectancy of less than two years.
5. Pregnancy -

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2014-06 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary function improvemnt | 6 months
  Clinical - COPD assessment test (CAT ) + lung volumes + diffusion capaciry and 6MWD .

CONTACTS AND LOCATIONS:
Overall Officials: david Stav, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Beer Yaakov, Israel